CLINICAL TRIAL: NCT01851122
Title: The Effect of the Amino Acid L-Theanine on Alertness and Vigilance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, David Bauer, Staff - Internal Medicine - Cardiology, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-GEN-11-0299
Record Dates: First submitted 2013-05-03; First posted 2013-05-10 (Estimated); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Theanine, (L)-Isomer
Keywords: l-theanine; alertness; well-being
MeSH Terms: interventions — theanine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo capsule (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo capsule
- L-theanine capsule (Experimental)
  Interventions: Dietary Supplement: L-theanine capsule

INTERVENTIONS:
Dietary Supplement: L-theanine capsule — L-theanine 250mg capsule
  Arms: L-theanine capsule
Dietary Supplement: Placebo capsule
  Arms: Placebo capsule

SUMMARY:
The amino acid l-theanine (the active ingredient in green tea) is considered to have a calming effect without causing sleepiness. This study evaluates whether l-theanine affects blood pressure, heart rate, alertness, and sense of well-being.

ELIGIBILITY:
Inclusion Criteria:

* adult
* able to swallow capsule

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Alertness | 48 hrs
  The average response time to identify a small rectangle shown on a computer screen.
Alertness | 48 hrs
  Degree of subjective alertness, measured on a visual analog scale
Well-Being | 48 hrs
  Sense of subjective well-being as measured on a visual analog scale

CONTACTS AND LOCATIONS:
Locations (1):
- Physicians at Sugar Creek, Sugar Land, Texas, United States